CLINICAL TRIAL: NCT06825923
Title: Precise Intervention of Obstructive Sleep Apnea Based on Phenotypic Characteristics and Endotypic Mechanisms
Brief Title: Precision OSA Therapy Based on Phenotypes and Endotypes
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Ding, Principal Investigator, Nanjing Medical University
Other Study IDs: 2025-SRFA-006
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; PALM; Phenotype; Endotype
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA Comprehensive Assessment Group: This group comprises patients diagnosed with Obstructive Sleep Apnea (OSA). Participants will undergo a comprehensive assessment that includes baseline demographic data collection, clinical symptom evaluation, polysomnography (PSG), Drug-Induced Sleep Endoscopy (DISE), and various physiological measurements to identify specific phenotypic and endotypic traits associated with OSA. This holistic evaluation aims to facilitate detailed phenotyping and generate predictive models for personalized treatment approaches.
  Interventions: Other: Clinical and Endotypic Assessmen

INTERVENTIONS:
Other: Clinical and Endotypic Assessmen — This observational study involves a detailed clinical and endotypic assessment of patients diagnosed with Obstructive Sleep Apnea (OSA). Assessments include polysomnography (PSG) to measure sleep patterns and disturbances, drug-induced sleep endoscopy (DISE) to evaluate upper airway obstruction, and various biomarker analyses to characterize endotypic traits. The study aims to collect comprehensive phenotypic and endotypic data to develop predictive models for OSA patient characterization and management.

SUMMARY:
Analyzing the phenotypic and endotypic characteristics of Sleep Apnea, along with DISE obstruction situations, is crucial for precise diagnosis and treatment. In this study, we aim to construct and apply a multidimensional predictive model based on four aspects: basic physiological characteristics of OSA, clinical phenotypes, mechanistic endotypes, and DISE obstruction levels. The study will begin by categorizing the clinical phenotypes; subsequently, it will quantify endotypic indicators based on PSG signal information and construct the PALM scale for Chinese individuals. Following this, a comprehensive clinical profile and a treatment efficacy prediction model for OSA patients will be built based on the results from the aforementioned multidimensional data.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is characterized by repeated episodes of upper airway obstruction and apneas during sleep, resulting in chronic intermittent hypoxemia, autonomic fluctuations, and sleep fragmentation. OSA is a heterogeneous disease influenced by multifactorial elements. The effectiveness of treatments and prognoses may vary due to differences in etiological factors, pathophysiological mechanisms, and clinical subtypes. Zinchuk et al. identified four clinical symptom and comorbidity-based subtypes and two subtypes based on polysomnography (PSG) indicators, which are useful for guiding treatment. However, relying solely on external phenotypes does not allow for analysis of intrinsic mechanisms, often leading to large treatment outcome disparities within the same phenotype due to different underlying mechanisms. Thus, the concept of OSA endotypes, which can elucidate pathophysiological mechanisms, has been introduced. OSA phenotypes are broadly defined as a classification of OSA patients related to clinically significant attributes such as symptoms, treatment response, underlying diseases, and quality of life; whereas endotypes refer to disease subtypes with distinct functional or pathophysiological mechanisms. There are at least four key pathophysiological endotypes in OSA, including 1) high upper airway closing pressure (Pcrit), 2) low arousal threshold (ArThr), 3) high loop gain (LG), and 4) impaired pharyngeal dilator muscle responsiveness. Each endotype represents a target or "treatable trait" from a mechanistic perspective. The advantages of OSA endotype quantification based on PSG signal information are evident. Eckert et al. proposed a potential classification of OSA patients into three subgroups based on the impairment of upper airway anatomy and the non-anatomical phenotypes (loop gain, arousal threshold, and muscle responsiveness) - the PALM scale. This phenotyping introduces different possible therapeutic strategies.

The same PSG outcomes may be caused by different endotypic mechanisms, and different endotypic mechanisms may lead to varying PSG outcomes, resulting in inconsistent treatment effects. To accurately align endotypes with PSG outcomes, a standard for obstruction anchoring is essential. Drug-induced sleep endoscopy (DISE) offers a bridge between the two by providing an assessment of the severity and plane of upper airway obstruction, which is related to both the severity of apneas and the upper airway closing pressure in the PALM model. In our preliminary research, the measurement of upper airway closing pressure and muscle responsiveness was achievable through DISE-PAP. Given the importance of distinguishing OSA patient phenotypic characteristics, quantifying endotypes, developing new indices, and assessing DISE obstruction planes, this study aims to construct and apply a multidimensional predictive model that integrates basic physiological characteristics of OSA, clinical phenotypes, mechanistic endotypes, and DISE obstruction planes. The study will start with the classification of clinical phenotypes, followed by the quantification of endotypic indicators based on PSG signal information and the construction of a PALM scale suitable for Chinese individuals. Subsequently, based on the results from the aforementioned multidimensional data, a comprehensive clinical portrait and predictive model of treatment outcomes for OSA patients will be built.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 80 years.
2. Diagnosed with Obstructive Sleep Apnea (OSA)(apnea-hypopnea index≥5/h).
3. First-time diagnosis, with no previous surgical interventions or CPAP treatment for OSA.
4. Ability and willingness to provide informed consent for participation in the study.

Exclusion Criteria:

1. History of severe stroke or cerebral hemorrhage, or presence of neurological or psychiatric conditions that could affect study results.
2. Presence of active malignancies or other severe underlying diseases, such as severe liver or kidney dysfunction. Diagnosed with diabetes or other significant vascular diseases.
3. Presence of severe chronic obstructive pulmonary disease (COPD), severe asthma, severe pulmonary hypertension, or heart failure caused by any condition.
4. Pregnancy or having other conditions that make participation in this study unsuitable.
5. Extremely debilitated patients or those with severe underlying conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve participants diagnosed with OSA who are not currently undergoing any active treatment for the condition. The study aims to explore the detailed phenotypic and endotypic characteristics of these patients to better understand OSA dynamics and develop predictive models for individualized treatment approaches.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Phenotype and Endotype Classification | 12 months post-enrollment.
  This outcome measure will evaluate the new phenotypic and endotypic features in OSA patients by integrating various clinical symptoms, traditional and novel PSG metrics, upper airway imaging indicators, diaphragm morphology and function parameters, and DISE results. A comprehensive classification system will be developed by combining these data points to classify OSA patients into distinct clinical phenotypes and endotypes. This classification aims to provide insights into the underlying pathophysiology of OSA and to better understand patient-specific characteristics for personalized treatment plans.
Multidimensional Predictive Model | End of the study, expected 24 months after enrollment.
  This outcome measure will assess the effectiveness of a multidimensional predictive model constructed using clinical phenotype, endotype, novel biomarkers, and DISE results. We used six commonly employed supervised machine learning algorithms: Random Forest, XGBoost, Support Vector Classifier (SVC), Logistic Regression, Multi-layer Perceptron (MLP), and Stacking Regression to classify OSA patients based on their survival status. The Stacking Regression model was designed by combining the outputs of Random Forest, XGBoost, and Support Vector Regression. The best-performing model will be selected to compute the final prediction, providing a powerful tool to predict the treatment response and clinical outcomes for OSA patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared. The informed consent will be ansigned before enrolled in the study and ensured to keep personal information confidential.

REFERENCES:
- [Background] Zinchuk A, Yaggi HK. Phenotypic Subtypes of OSA: A Challenge and Opportunity for Precision Medicine. Chest. 2020 Feb;157(2):403-420. doi: 10.1016/j.chest.2019.09.002. Epub 2019 Sep 17. PMID 31539538
- [Background] Zinchuk AV, Gentry MJ, Concato J, Yaggi HK. Phenotypes in obstructive sleep apnea: A definition, examples and evolution of approaches. Sleep Med Rev. 2017 Oct;35:113-123. doi: 10.1016/j.smrv.2016.10.002. Epub 2016 Oct 12. PMID 27815038
- [Background] Aishah A, Eckert DJ. Phenotypic approach to pharmacotherapy in the management of obstructive sleep apnoea. Curr Opin Pulm Med. 2019 Nov;25(6):594-601. doi: 10.1097/MCP.0000000000000628. PMID 31503212
- [Background] Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med. 2013 Oct 15;188(8):996-1004. doi: 10.1164/rccm.201303-0448OC. PMID 23721582
- [Background] Eckert DJ. Phenotypic approaches to obstructive sleep apnoea - New pathways for targeted therapy. Sleep Med Rev. 2018 Feb;37:45-59. doi: 10.1016/j.smrv.2016.12.003. Epub 2016 Dec 18. PMID 28110857
- [Background] Van den Bossche K, Van de Perck E, Kazemeini E, Willemen M, Van de Heyning PH, Verbraecken J, Op de Beeck S, Vanderveken OM. Natural sleep endoscopy in obstructive sleep apnea: A systematic review. Sleep Med Rev. 2021 Dec;60:101534. doi: 10.1016/j.smrv.2021.101534. Epub 2021 Aug 3. PMID 34418668